CLINICAL TRIAL: NCT01437358
Title: Epidural Analgesia in Intensive Care Unit Patients: an Observational Prospective Multicenter Feasibility and Safety Study
Brief Title: Epidural Analgesia in Intensive Care Unit (APD-REA: Analgesie PeriDurale en REAnimation)
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0100
Record Dates: First submitted 2011-08-30; First posted 2011-09-20 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Critical Illness; Epidural Analgesia
Keywords: Epidural catheter; Epidural analgesia; Intensive care unit; Safety
MeSH Terms: conditions — Critical Illness | interventions — Analgesia, Epidural

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- intensive care unit
  Interventions: Other: Epidural analgesia

INTERVENTIONS:
Other: Epidural analgesia — The purpose of this observational prospective study is to describe the safety and feasibility of this analgesia technique in ICU patients

SUMMARY:
Epidural analgesia (EA) has been mainly investigated during the perioperative period. In the intensive care unit settings, EA should be proposed in critically ill patients, such as postoperative or trauma patients, typically. Recent findings also support anti-inflammatory, vascular or respiratory effects for EA, beyond its analgesic effects. However, data on EA safety and feasibility in the intensive care unit settings are still lacking. The purpose of this observational prospective study is to describe the safety and feasibility of this analgesia technique in ICU patients.

DETAILED DESCRIPTION:
BACKGROUND:

Epidural analgesia (EA) has been mainly investigated during the perioperative period. In the intensive care unit settings, EA should be proposed in critically ill patients, such as postoperative or trauma patients, typically. Recent findings also support anti-inflammatory, vascular or respiratory effects for EA, beyond its analgesic effects. However, data on EA safety and feasibility in the intensive care unit settings are still lacking.

DESIGN NARRATIVE:

This observational multicenter prospective clinical study will report the incidence of EA-related complications, such as infectious or neurologic complications, and the mean duration of EA in the ICU settings.

Patients admitted in three intensive care units (two from an University Hospital and one from a local hospital) and receiving EA will be included in the study, whether the EA catheter is inserted in the ICU or outside the ICU, e.g. in the operating room. Demographics, clinical and biological data will be recorded prospectively. The main goal is to evaluate the safety and feasibility of EA in critically ill patients, being assumed this technique is currently and routinely used in our intensive care units, in accordance with national and international guidelines on epidural analgesia practice.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring epidural analgesia, whether the epidural analgesia catheter is inserted in the ICU or outside the ICU, e.g. in the operating room.

Exclusion Criteria:

* none (besides classic contra-indications for epidural analgesia catheter insertion, e.g. coagulation disorder, local infection…)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring epidural analgesia, whether the epidural analgesia catheter is inserted in the ICU or outside the ICU, e.g. in the operating room
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of epidural analgesia-related complications | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand; Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand; Russel CHABANNE, Principal Investigator — University Hospital, Clermont-Ferrand; Bernard CLAUD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Chabanne R, Sossou A, Bertrand PM, Kauffmann S, Chartier C, Guerin R, Imhoff E, Zanre L, Brenas F, Bazin JE, Constantin JM. Epidural analgesia in the intensive care unit: An observational series of 121 patients. Anaesth Crit Care Pain Med. 2015 Aug;34(4):217-23. doi: 10.1016/j.accpm.2014.12.002. Epub 2015 May 23. PMID 26004880